CLINICAL TRIAL: NCT05801770
Title: An Observational Medical Trial Assessing Patterns in Experiences of Participants of Head and Neck Cancer Clinical Trials
Brief Title: Discovering Factors in Head and Neck Cancer Patients' Clinical Study Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80513342
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enrollment in clinical trials usually favors a particular demographic group. But there is limited research available to explain what study attributes affect the completion of these specific demographic groups.

This trial will evaluate the safety and efficacy of head and neck cancer treatments. The focus will be on tracking the rates of completion and withdrawal among these individuals.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future head and neck cancer studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is able and willing to comply with the treatment/follow-up schedule and requirements
* Patient must provide written informed consent

Exclusion Criteria:

* Participants who are vulnerable to any intervention
* Women who are pregnant, intend to become pregnant, or are lactating
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational head and neck cancer clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a clinical study. | 3 months
Number of study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaanders JHAM, van den Bosch S, Kleijnen J. Comparison of Patients With Head and Neck Cancer in Randomized Clinical Trials and Clinical Practice: A Systematic Review. JAMA Otolaryngol Head Neck Surg. 2022 Jul 1;148(7):670-676. doi: 10.1001/jamaoto.2022.0890. PMID 35587353
- [Background] Simon C, Caballero C. Quality Assurance and Improvement in Head and Neck Cancer Surgery: From Clinical Trials to National Healthcare Initiatives. Curr Treat Options Oncol. 2018 May 24;19(7):34. doi: 10.1007/s11864-018-0552-y. PMID 29797284
- [Background] Argiris A, Karamouzis MV, Raben D, Ferris RL. Head and neck cancer. Lancet. 2008 May 17;371(9625):1695-709. doi: 10.1016/S0140-6736(08)60728-X. PMID 18486742

DOCUMENTS (1):
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT05801770/ICF_000.pdf